CLINICAL TRIAL: NCT00535366
Title: A Randomised, Phase II, Double-Blind, Double-Dummy, Four-period Crossover Efficacy and Safety Comparison of 4-Week Treatment Periods of Blinded Fluticasone (500 mcg Bid, MDI), Ciclesonide (400 mcg qd, MDI), Ciclesonide (800 mcg qd, MDI) or Placebo in Free Combination With Open-Label Tiotropium (18 mcg qd, HandiHaler) and Salmeterol (50 mcg Bid, Diskus) in Patients With COPD.
Brief Title: Efficacy and Safety Comparison of Steroid or Placebo in Combination With Salmeterol and Tiotropium in COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1249.1; Eudract2007-003169-42
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate; Fluticasone

ARMS (4):
- Tiotropium+salmeterol+fluticasone (Experimental)
  Interventions: Drug: Tiotropium; Drug: Salmeterol; Drug: Fluticasone
- Tiotropium+salmeterol+ciclesonide low (Experimental)
  Interventions: Drug: Tiotropium; Drug: Salmeterol; Drug: Ciclesonide low
- Tiotropium+salmeterol+ciclesonide high (Experimental)
  Interventions: Drug: Tiotropium; Drug: Salmeterol; Drug: Ciclesonide high
- Placebo (Placebo Comparator)
  Interventions: Drug: Tiotropium; Drug: Salmeterol; Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium — Oral inhalation by HandiHaler® device
Drug: Salmeterol — Oral inhalation from Diskus®
Drug: Fluticasone — Oral inhalation from metered dose inhaler (MDI)
  Arms: Tiotropium+salmeterol+fluticasone
Drug: Ciclesonide low — Oral inhalation from MDI
  Arms: Tiotropium+salmeterol+ciclesonide low
Drug: Ciclesonide high — Oral inhalation from MDI
  Arms: Tiotropium+salmeterol+ciclesonide high
Drug: Placebo — Oral inhalation from MDI
  Arms: Placebo

SUMMARY:
This efficacy and safety study compares four different combinations of blinded inhaled steroid treatments on top of open-label tiotropium and salmeterol in patients with chronic obstructive pulmonary disease (COPD). The primary objective is the effect on lung function parameters.

ELIGIBILITY:
Inclusion Criteria:

* Relatively stable, moderate to severe COPD
* Male or female patients 40 years of age or older.
* Current or ex-smokers with a smoking history of more than 10 pack years

Exclusion Criteria:

* Other significant disease that can influence the study results or be a safety risk for the patient
* Other medication that can influence the study results
* Hypersensitivity to the study medication
* Patients with unstable COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Trough FEV1 response at the end of each 4 week period of randomised treatment | 4 weeks

SECONDARY OUTCOMES:
Trough forced vital capacity (FVC) response after 4 weeks of each blinded treatment | after 4 weeks of each blinded treatment
All adverse events | 24 weeks
Pulse rate and blood pressure (seated) | 24 weeks
FEV1 and FVC morning peak response | day 1 and day 28 of each blinded treatment
FEV1 and FVC evening peak response | day 1 and day 28 of each blinded treatment
FEV1 AUC (0-3h), after 4 weeks of each blinded treatment | after 4 weeks of each blinded treatment
FEV1 AUC (12-15h) after 4 weeks of each blinded treatment | after 4 weeks of each blinded treatment
FVC AUC (0-3h) after 4 weeks of each blinded treatment | after 4 weeks of each blinded treatment
FVC AUC (12-15h) after 4 weeks of each blinded treatment | after 4 weeks of each blinded treatment
Trough and peak inspiratory capacity (IC) and vital capacity (VC) response in the morning of day 1 and at day 28 of each treatment period | day 1 and day 28 of each blinded treatment
Weekly mean pre-dose morning and evening peak expiratory flow (PEF) | 28 weeks
Weekly mean number of occasions of rescue therapy used per day | 28 weeks
Mahler Dyspnea Indices (TDI) collected at the end of each treatment period and each wash-out period | 28 weeks
Fractional exhaled nitric oxide after 4 weeks of each blinded treatment | after 4 weeks of each blinded treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- Belgium (4):
  - 1249.1.32003 Boehringer Ingelheim Investigational Site, Genk
  - 1249.1.32001 Boehringer Ingelheim Investigational Site, Ghent
  - 1249.1.32002 Boehringer Ingelheim Investigational Site, Hasselt
  - 1249.1.32004 Boehringer Ingelheim Investigational Site, Ostend
- 1249.1.45001 Boehringer Ingelheim Investigational Site, Aarhus C, Denmark
- Germany (3):
  - 1249.1.49001 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1249.1.49002 Boehringer Ingelheim Investigational Site, Mannheim
  - 1249.1.49003 Boehringer Ingelheim Investigational Site, Weinheim
- Netherlands (4):
  - 1249.1.31002 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1249.1.31003 Boehringer Ingelheim Investigational Site, Harderwijk
  - 1249.1.31001 Boehringer Ingelheim Investigational Site, Heerlen
  - 1249.1.31004 Boehringer Ingelheim Investigational Site, Veldhoven